CLINICAL TRIAL: NCT00201773
Title: A Phase II Trial of Exemestane (Aromasin) in Combination With Celecoxib (Celebrex) as Neoadjuvant Treatment in Postmenopausal Women With Stage II, III, and IV Breast Cancer
Brief Title: Exemestane With Celecoxib as Neoadjuvant Treatment in Postmenopausal Women With Stage II, III, and IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Stephen Povoski, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0245
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: Post-Menopause; Neoadjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Celecoxib; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exemestane & Celecoxib (Experimental): Patients will receive exemestane 25 mg orally per day for 8 weeks. Starting in the 9th week, patients will receive celecoxib 400 mg orally twice per day for 8 weeks in addition to exemestane.
  Interventions: Drug: Exemestane; Drug: Celecoxib; Other: Correlative studies

INTERVENTIONS:
Drug: Exemestane — 25 mg orally once per day for 16 weeks.
  Other Names: Aromasin
Drug: Celecoxib — given orally at two 200 mg capsules (400 mg) twice per day. Patients assigned to receive 400 mg twice per day should be instructed to take the drug with food.
  Other Names: Celebrex
Other: Correlative studies
  Other Names: biopsy; tissue specimens; tissue samples

SUMMARY:
To test whether the addition of the COX-2 inhibitor, celecoxib, will decrease the gene expression of CYP19 in breast cancers collected from postmenopausal women that receive neoadjuvant exemestane.

DETAILED DESCRIPTION:
Rationale: In postmenopausal women, the main source of estrogen is through the conversion of androgens, or sex hormones produced by the adrenal glands. An enzyme called aromatase carries out this process. Exemestane, an aromatase inhibitor, blocks production of estrogens. Research indicates that the gene responsible for aromatase activity is CYPO19. Therefore, exemestane helps to inhibit aromatase activity through CYP019. Along with CYP019, another gene associated with breast cancer is an overexpression of COX-2 enzymes. Research suggests that COX-2 overexpression can cause cancer cell division, increased blood flow to tumors, and metastases. Celecoxib blocks COX-2 activity and produces fewer side effects compared with other non-steroidal inflammatory drugs (NSAIDs). This study builds on previous research to test the combination of exemestane and celecoxib for breast cancer.

Purpose: This study is evaluating the safety and efficacy of exemestane and celecoxib before surgery for stage II, III, and IV breast cancer in postmenopausal women. Tests will analyze the CYP019 gene after these treatments.

Treatment: Patients in this study will receive exemestane and celecoxib. Both drugs will be given to patients as oral pills. Exemestane will be taken daily for sixteen weeks. Starting in week 9, celecoxib will be taken twice daily for eight weeks. Therefore, during weeks 9-16, patients will be taking both exemestane and celecoxib. Several tests and exams will be given throughout the study to closely monitor patients, including a biopsy performed after the first 8 weeks on exemestane. After sixteen weeks on exemestane and celecoxib, patients will have breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Must be female with histologically confirmed breast cancer
* Stage II-IV disease
* ER and/or PR positive
* ECOG Performance Status 0-1
* Tumor must be present following core needle biopsy as determined by physical exam or radiographic evaluation.
* Postmenopausal
* No prior treatment for current breast cancer. No other active malignancy is allowed.Adequately treated basal cell, squamous cell skin cancer, in situ cervical cancer, or any other cancer from which the patient has been disease-free for 5 years is permitted. Biphosphonates and palliative radiation for bone metastasis is permitted while on study.
* Hormone replacement therapy must be discontinued. It is not permitted during the time on study.

Exclusion Criteria:

* Known history of aspirin or NSAID induced asthma, urticaria or allergic reactions; or allergy to sulfonamides severe enough in nature to require emergency room treatment or hospitalization.
* History of myocardial infarction or other thrombotic events.
* Inflammatory breast cancer (edema or ulceration of the skin of the breast).
* Significant renal dysfunction (serum creatinine > 1.5 x upper limit of normal).
* Significant hepatic dysfunction (serum bilirubin > 1.5 x upper limit of normal or AST, ALT > 3 x upper limit of normal)
* ANC <1.5, platelets <100,000 K/uL, and hemoglobin < 9 g/dL.
* Use of other COX-2 inhibitors such as rofecoxib (Vioxx®, aspirin, trisalicylate (Trilisate®), is not permitted during the time on study. No washout period is required. Baby aspirin, 81 mg po daily, is permitted.
* Use of NSAID's such as ibuprofen (Advil® or Motrin®), naproxyn (Aleve® Naprosyn®, or Anaprox®), etodolac (Lodine®), oxaprozin (Daypro®), difusanil (Dolobid®), nabumetone (Relafin®), or tolmetin (Tolectin®) is not permitted during the time on study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-07; Primary Completion 2007-11 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Povoski, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of postmenopausal women between January 2003 and July 2007
Groups:
- Exemestane & Celecoxib: Patients will receive exemestane 25 mg orally per day for 8 weeks. Starting in the 9th week, patients will receive celecoxib 400 mg orally twice per day for 8 weeks in addition to exemestane.
  Exemestane: 25 mg orally once per day for 16 weeks.
  Celecoxib: given orally at two 200 mg capsules (400 mg) twice per day. Patients assigned to receive 400 mg twice per day should be instructed to take the drug with food.
  Correlative studies
Period: Overall Study
Arm/Group | Exemestane & Celecoxib
Started | 22
Completed 8 Weeks of Planned Therapy | 16
Received All Exemestane Therapy | 5
Stopped Exemestane After 4 Weeks | 1
Completed | 16
Not Completed | 6

BASELINE CHARACTERISTICS:
Groups:
- Exemestane & Celecoxib: Patients will received exemestane 25 mg orally per day for 8 weeks. Starting in the 9th week, patients will receive celecoxib 400 mg orally twice per day for 8 weeks in addition to exemestane.
  Exemestane: 25 mg orally once per day for 16 weeks.
  Celecoxib: given orally at two 200 mg capsules (400 mg) twice per day. Patients assigned to receive 400 mg twice per day and instructed to take the drug with food.
  Correlative studies
Arm/Group | Exemestane & Celecoxib
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 63 [49 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Region of Enrollment [Number; unit: patients]
  United States | 22
ECOG (Eastern Cooperative Oncology Group) Performance Status 0-1 [Number; unit: patients] — ECOG Performance Status 0 is defined as fully active, able to carry on all pre-disease performance without restriction.
  ECOG Performance Status1 is defined as restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  patients | 22
Menopause Status of Postmenopausal [Number; unit: patients] | 22
Progesterone Receptor status [Number; unit: patients]
  Positive | 16
  Negative | 6
Her-2 FISH [Number; unit: patients] — Fluorescence in situ hybridization
  patients
    Positive | 4
    Negative | 8
    Not available | 10
Histology [Number; unit: patients]
  Invasive | 15
  Lobular | 5
  Mixed invasive and lobular | 2
Clinical Axillary Status [Number; unit: patients]
  Positive | 7
  Negative | 15
Axillary Nodal Evaluation [Number; unit: patients]
  Fine needle aspiration | 2
  Sentinel | 1
Clinical Stage [Number; unit: patients]
  I (cancer cells confined to limited area) | 1
  IIA (evidence cancer has begun to grow/spread) | 14
  IIB (tumor between 2-5 cm or larger) | 3
  IIIA (cancer considered advanced) | 3
  Occult primary (axillary metastases) | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Decreased Gene Expression of CYP19 in Breast Cancer by Adding COX-2 Inhibitor to Exemestane
Description: Collected from postmenopausal women that receive neoadjuvant exemestane.
Time Frame: up to 16 weeks
Population: Comparison of immunohistochemistry (IHC) Allred Differences with Neoadjuvant Therapy
Measure: Number; unit: patients
Groups:
- Exemestane + Celecoxib: Exemestane + celecoxib (16 weeks) vs. Baseline
- Exemestane: Exemestane (8 weeks) vs. Baseline
Arm/Group | Exemestane + Celecoxib | Exemestane
Number analyzed (Participants) | 14 | 9
patients | 0 | 0

2. Secondary Outcome: Evaluate Response Rate of Neoadjuvant Exemestane and Celecoxib in Postmenopausal Women.
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response, Disappearance of all target lesions; Partial Response, >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease, <30% decrease in the sum of the longest diameter of target lesions; Progressive Disease, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: up to 16 weeks
Population: Clinical Response was determined by physical exam and breast Ultrasound at baseline and repeated at 8 weeks and 16 weeks, and pathological response by histopathological examination of primary tumor and axillary nodes after definitive breast cancer surgery.
Measure: Number; unit: patients
Arm/Group | Exemestane & Celecoxib
Number analyzed (Participants) | 22
patients
  Complete Response | 0
  Partial Response | 5
  Stable Disease | 1
  Progressive Disease | 1
  Non-measurable | 15

ADVERSE EVENTS:
Description: Toxicities were graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. The same patient could be counted more than once if the same toxicity occured during treatment with exemestane alone and again when exemestane was combined with celecoxib.
Groups:
- Exemestane Alone; Exemestane + Celecoxib: Patients will receive exemestane 25 mg orally per day for 8 weeks. Starting in the 9th week, patients will receive celecoxib 400 mg orally twice per day for 8 weeks in addition to exemestane.
  Exemestane: 25 mg orally once per day for 16 weeks.
  Celecoxib: given orally at two 200 mg capsules (400 mg) twice per day. Patients assigned to receive 400 mg twice per day should be instructed to take the drug with food.
Arm/Group | Exemestane Alone | Exemestane + Celecoxib
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 22/22 | 22/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exemestane Alone (N=22) | Exemestane + Celecoxib (N=22)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 5 (5)
Heartburn (Gastrointestinal disorders) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 5 (5)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 10 (10) | 6 (6)
Hot Flashes (Vascular disorders) | 9 (9) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Edema (Vascular disorders) | 0 (0) | 2 (2)
Renal Insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 4 (4)
Sensory Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Lower Gastrointestional Bleed (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes